CLINICAL TRIAL: NCT05202145
Title: A Three-Part Phase 1 Study to Evaluate the Potential Drug Interactions Between ALXN2050 and Cyclosporine, Tacrolimus, and Mycophenolate Mofetil in Healthy Adult Participants
Brief Title: Drug-Drug Interaction (DDI) Study of ALXN2050 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN2050-HV-110
Record Dates: First submitted 2022-01-10; First posted 2022-01-21 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: ALXN2050; Cyclosporine; Tacrolimus; Mycophenolate Mofetil; Drug-Drug Interaction; Pharmacokinetics; Safety; Factor D Inhibitor
MeSH Terms: interventions — rhoA GTP-Binding Protein; Cyclosporine; Tacrolimus

STUDY DESIGN:
Intervention Model Description: This will be a 3-part study with each part being an open-label, fixed-sequence study in healthy adult participants. The 3 parts of the study may be conducted concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - Cyclosporine (Experimental): Participants will receive ALXN2050 and cyclosporine in a fixed sequence over 3 periods.
  Period 1: Participants will receive multiple doses of ALXN2050.
  Period 2: Participants will receive multiple doses of cyclosporine.
  Period 3: Participants will receive multiple doses of ALXN2050 co-administered with multiple doses of cyclosporine.
  There will be a washout period between the last dose of ALXN2050 in Period 1 and the first dose of cyclosporine in Period 2 and between the last dose of cyclosporine in Period 2 and the first dosing in Period 3.
  Interventions: Drug: ALXN2050; Drug: Cyclosporine
- Part 2 - Tacrolimus (Experimental): Participants will receive tacrolimus and ALXN2050 in a fixed sequence over 2 periods.
  Period 1: Participants will receive a single dose of tacrolimus.
  Period 2: Participants will receive multiple doses of ALXN2050 alone and co-administered with a single dose of tacrolimus.
  There will be a washout period between the dose of tacrolimus in Period 1 and the first dose of ALXN2050 in Period 2.
  Interventions: Drug: ALXN2050; Drug: Tacrolimus
- Part 3 - MMF (Experimental): Participants will receive MMF and ALXN2050 in a fixed sequence over 2 periods.
  Period 1: Participants will receive a single dose of MMF.
  Period 2: Participants will receive multiple doses of ALXN2050 alone and co-administered with a single dose of MMF.
  There will be a washout period between the dose of MMF in Period 1 and the first dose of ALXN2050 in Period 2.
  Interventions: Drug: ALXN2050; Drug: MMF

INTERVENTIONS:
Drug: ALXN2050 — Oral tablet.
  Other Names: ACH-0145228 (formerly)
Drug: Cyclosporine — Oral capsule.
  Arms: Part 1 - Cyclosporine
Drug: Tacrolimus — Oral capsule.
  Arms: Part 2 - Tacrolimus
Drug: MMF — Oral tablet.
  Arms: Part 3 - MMF

SUMMARY:
This study will evaluate the potential drug interactions between ALXN2050 and cyclosporine (Part 1), between ALXN2050 and tacrolimus (Part 2), and between ALXN2050 and mycophenolate mofetil (MMF) (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy with no clinically significant or relevant abnormalities as determined by medical history, physical or neurological examination, vital signs, 12-lead electrocardiogram, screening clinical laboratory profiles (hematology, biochemistry, coagulation, and urinalysis), as deemed by the Investigator or designee at Screening.
* Body mass index within the range 18.0 to 32.0 kilograms (kg)/meter^2, inclusive, with a minimum body weight of 50.0 kg at Screening.

Exclusion Criteria:

* History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
* Participation in another investigational drug or investigational device study within 5 half- lives (if known) or 30 days prior to the first dose of study intervention, whichever is longer.
* History of drug or alcohol abuse within 2 years prior to the first dose of study intervention or positive drugs-of-abuse or alcohol screen at Screening or Day -1; current tobacco users or smokers or a positive cotinine test at Screening.
* Donation of whole blood from 3 months prior to the first dose of study intervention, or of plasma from 30 days prior to the first dose of study intervention; receipt of blood products within 6 months prior to the first dose of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Part 1 Cyclosporine: Area Under The Concentration-Time Curve From Time Zero To The 12-hour Time Point (AUC0-12) Following Multiple Dose Cyclosporine Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose
Part 1: ALXN2050 AUC0-12 Following Multiple Dose ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Cyclosporine | Up to 72 hours postdose
Part 1: Cyclosporine Maximum Observed Concentration (Cmax) Following Multiple Dose Cyclosporine When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose
Part 1: ALXN2050 Cmax Following Multiple Dose ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Cyclosporine | Up to 72 hours postdose
Part 1: Cyclosporine Time To Maximum Plasma Concentration (Tmax) Following Multiple Dose Cyclosporine When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose
Part 1: ALXN2050 Tmax Following Multiple Dose ALXN2050 When Dosed Alone Versus When Dosed In The Presence Of Steady-state Cyclosporine | Up to 72 hours postdose
Part 2: Tacrolimus Area Under The Concentration-Time Curve From Time Zero To The Last Observed Concentration (AUC0-t) Following Single Dose Tacrolimus When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 144 hours postdose
Part 2: Tacrolimus Area Under the Concentration-Time Curve From Time Zero To Infinity (AUC0-inf) Following Single Dose Tacrolimus When Dosed Alone Versus When Dosed In The Presence of Steady-state ALXN2050 | Up to 144 hours postdose
Part 2: Tacrolimus Cmax Following Single Dose Tacrolimus When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 144 hours postdose
Part 2: Tacrolimus Tmax Following Single Dose Tacrolimus When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 144 hours postdose
Part 3: Mycophenolic Acid (MPA) And Mycophenolic Acid Glucuronide (MPAG) (Active Metabolites Of MMF) AUC0-t Following Single Dose MMF When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose
Part 3: MPA and MPAG AUC0-inf Following Single Dose MMF When Dosed Alone Versus When Dosed In The Presence Of Steady-State ALXN2050 | Up to 72 hours postdose
Part 3: MPA And MPAG Cmax Following Single Dose MMF When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose
Part 3: MPA And MPAG Tmax Following Single Dose MMF When Dosed Alone Versus When Dosed In The Presence Of Steady-state ALXN2050 | Up to 72 hours postdose

SECONDARY OUTCOMES:
Parts 1-3: Number of Participants Experiencing Treatment-emergent Adverse Events | Day 1 through up to 12 days postdose

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR